CLINICAL TRIAL: NCT01140568
Title: A Phase II Study of PDGFR Kinase Inhibitor in Biomarker-Enriched Recurrent Malignant Gliomas
Brief Title: Study of Platelet Derived Growth Factor Receptor (PDGFR) in Recurrent Malignant Gliomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: David Piccioni, M.D., Ph.D (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, David Piccioni, M.D., Ph.D, Assistant Clinical Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 091728
Record Dates: First submitted 2010-06-08; First posted 2010-06-09 (Estimated); Results first posted 2020-04-24 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Glioma
Keywords: glioma; PDGFR; kinase; inhibitor; malignant; nilotinib
MeSH Terms: conditions — Glioma | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- nilotinib (Experimental): Patients will take nilotinib twice daily at the standard dose of 400mg taken by mouth twice a day until disease progression or development of unacceptable side effects.
  Interventions: Drug: nilotinib

INTERVENTIONS:
Drug: nilotinib — 400mg po (orally) BID (twice daily)
  Other Names: Tasigna

SUMMARY:
The purpose of this study is to determine the survival, disease response, and side effects of Tasigna® (nilotinib) in patients who have malignant gliomas and are positive for Platelet Derived Growth Factor Receptor (PDGFR) amplification. This study is designed to test the hypothesis that patients with malignant gliomas with PDGFR amplification are sensitive to PDGFR kinase inhibitors.

DETAILED DESCRIPTION:
Malignant gliomas (MG), including anaplastic gliomas (AG) and glioblastoma (GBM), are the most common primary brain tumor. Standard of care (surgery, radiotherapy, and temozolomide at initial diagnosis) results in a median survival of only 14 months. For patients with recurrent disease, conventional chemotherapy is generally ineffective with response rates <20%. Clearly there is need for improved treatments. Recent genome-wide studies have confirmed that GBM is a heterogeneous group of diseases that can be subclassified by shared genetic aberrations. The implication is that, in part, the underlying genetics may determine responsiveness to treatments and thus allow us to personalize therapy.

This is an, open-label, non-randomized, phase II study with oral nilotinib in adult patients with biomarker-enriched, recurrent malignant gliomas who have developed tumor progression after standard therapy. Patients will be treated with oral nilotinib (starting with the labeled dose of 400 mg) daily until disease progression or intolerance. One cycle is defined as 28 days.

Approximately 50 evaluable patients will be enrolled in this study, with 32 (grade IV) and 18 (grade III) in separate arms.

All patients will undergo clinical evaluation after each 28-day cycle. Neuroimaging studies (MRI) will be performed at baseline, 4 weeks, 8 weeks and then after every 2 cycles (8 weeks). If a contraindication for MRI's exists, patients will undergo contrast-enhanced CT scans. Laboratory tests will be obtained weekly during the first 4 weeks, and then on days 1 and 15 of all subsequent cycles. Patients will remain on study medication unless they develop tumor progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent prior to participation in the study and any related procedures being performed.
* Participants must have agreed to and signed an authorization for the release of their protected health information.
* Subjects must be able to adhere to the dosing and visit schedules, and agree to record medication times accurately and consistently in a daily diary.
* Participants must have a life expectancy of at least 8 weeks.
* Patients greater than 18 years of age.
* Histologically documented diagnosis of proven glioblastoma (GBM), or anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO), and anaplastic mixed oligoastrocytoma (AMO). Patients are eligible if the original local pathology was lower-grade glioma. Pathology will be read centrally to confirm diagnosis.
* Documentation of amplified PDGFRA by fluorescent in-situ hybridization (FISH), colorimetric in-situ hybridization (CISH), or quantitative PCR from tumor tissue (=>3 copy number). Availability of unstained paraffin slides or the paraffin block of pretreatment baseline tissue is required for eligibility and for molecular analysis and would help to identify molecular predictors of outcome (all patients).
* Participants must have a Karnofsky Performance Status (KPS) ≥ 60.
* Adequate end organ function, defined as the following:

  * Hematology:

    * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
    * Platelet count ≥ 100 x 109/L
    * Hemoglobin ≥ 9.0 g/dL
    * White blood cell (WBC) count ≥ 3.0 x 109/L
  * Biochemistry:

    * AST/SGOT and ALT/SGPT ≤ 2.5 x institution's ULN
    * Total bilirubin ≤ 1.5 x institution's ULN
    * Serum creatinine ≤ 1.5 x institution's ULN or 24-hour creatinine clearance ≥ 50 ml/min
    * Alkaline phosphatase (ALP) ≤ 2.5 x ULN unless considered tumor related
* Patients must have the following laboratory values within normal limits (WNL) at the local institution lab or corrected to WNL with supplements prior to first dose of study medication.

  * Potassium (WNL)
  * Magnesium (WNL)
  * Phosphorous (WNL)
  * Calcium (WNL)
  * Coagulation studies:

    * INR < 1.5
    * PTT within institution's normal range, unless receiving therapeutic low molecular weight heparin
* Female patients of childbearing potential must have negative pregnancy test within 7 days before initiation of study drug dosing. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male and female patients of reproductive potential must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug.
* Participants must have an unequivocal progression by magnetic resonance imaging (MRI) or computed tomography (CT) scan. A scan must be performed within 14 days prior to registration and on a steroid dose that has been stable for at least 5 days. If the steroid dose is increased between the date of imaging and registration, a new baseline MRI/CT is required. The same type of scan, i.e., MRI or CT must be used throughout the period of protocol treatment for tumor measurement. A patient who develops a contraindication to undergo an MRI scan during study treatment may remain on study and undergo contrast enhanced CT scans.
* Patients must have failed prior radiation therapy and must have an interval of greater than or equal to 60 days from the completion of radiation therapy to study entry.
* Subjects must have recovered from the toxic effects of prior therapy. Residual toxicity from any previous treatment must be ≤ Grade 1.
* Patients must have sufficient time for recovery from prior therapy: 28 days from any investigational agent, 28 days from prior cytotoxic therapy (except 23 days from prior temozolomide, 14 days from vincristine, 42 days from nitrosoureas, 21 days from procarbazine administration), and 7 days for non-cytotoxic agents, e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc. (radiosensitizer does not count).
* Patients with prior therapy that included interstitial brachytherapy or stereotactic radiosurgery must have confirmation of true progressive disease rather than radiation necrosis based upon positron emission tomography (PET), Thallium scanning, MR spectroscopy or surgical documentation of disease.
* Subjects who have undergone recent resection of recurrent or progressive tumor will be eligible as long as all of the following conditions apply:

  * Prior to initiating therapy, 4 weeks must have elapsed since surgery;
  * Subjects must have recovered from surgical-related trauma;
  * Wound healing needs to have occurred.

Exclusion Criteria:

* Patients who received PDGFR inhibitors (imatinib, sunitinib, nilotinib, etc.) previously are excluded (patients who received PDGFR antibody based treatment however are allowed).
* History of intratumoral or peritumoral hemorrhage if deemed significant by the treating physician.
* For patients requiring anticoagulation therapy, only therapeutic low molecular weight heparin or factor Xa inhibitors are permitted.
* Due to the potential interaction between nilotinib and enzyme-inducing anti-epileptic drugs (EIAED), only patients on non-enzyme inducing anti-epileptic drugs (NEIAED) or on no anti-epileptic drugs are eligible.
* Patient is < 3 years free of another primary malignancy except: if the other primary malignancy is not currently clinically neither significant nor requiring active intervention, or if other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ. Existence of any other malignant disease is not allowed.
* Female patients who are pregnant or breast-feeding, or intends to become pregnant during the study.
* Any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy.
* Patient has a rare hereditary problem of galactose intolerance, severe lactase deficiency or of glucose-galactose malabsorption.
* Patients with any disease that will obscure toxicity or dangerously alter drug metabolism.
* Patient with electrolyte abnormality (e.g., hypokalemia, hypomagnesemia, hypophosphatemia, hyperkalemia, hypocalcemia, hyponatremia) unless the level can be corrected to normal levels prior to initiating study drug.
* Patient has a known diagnosis of human immunodeficiency virus (HIV) infection.
* Patient received chemotherapy within 4 weeks (6 weeks for nitrosourea) prior to study entry, unless the disease is rapidly progressing.
* Concomitant use of any anti-cancer therapy or radiation therapy, or any other investigational agent.
* Impaired cardiac function including any of the following:

  * Congenital long QT syndrome or a known family history of long QT syndrome;
  * History or presence of clinically significant ventricular or atrial tachyarrhythmias
  * Clinically significant resting bradycardia (< 50 beats per minute)
  * Inability to monitor the QT interval by ECG
  * QTc > 450 msec on baseline ECG. If QTc > 450 and electrolytes are not within normal ranges, electrolytes should be corrected and then the patient re-screened for QTc
  * Myocardial infarction within 1 year of starting study drug
  * Other clinically significant heart disease (e.g., unstable angina, congestive heart failure, or uncontrolled hypertension)
* Patients currently receiving treatment with strong CYP3A4 inhibitors and treatment cannot be either discontinued or switched to a different medication prior to starting study drug. See link for complete list of CYP3A4 inhibitors (http://medicine.iupui.edu/clinpharm/ddis/table.asp)
* Patient currently receiving treatment with any medications that have the potential to prolong the QT interval and cannot be either discontinued or switched to a different medication prior to starting study drug. See link for a comprehensive list of agents that prolong the QT interval (http://www.azcert.org/medical-pros/drug-lists/printable-drug-list.cfm).
* Impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection or gastric bypass surgery).
* Acute or chronic pancreatic disease.
* Another malignancy that is clinically significant or requires active intervention (chemotherapy or radiation)
* Severe or uncontrolled medical conditions (i.e., uncontrolled diabetes, active or uncontrolled infection).
* Acute or chronic liver or severe renal disease
* History of significant congenital or acquired bleeding disorder.
* Major surgery within 4 weeks prior to Day 1 of study or who have not recovered from prior surgery.
* Treatment with other investigational agents within 30 days of Day 1.
* History of non-compliance to medical regimens or inability to grant consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-04-21 (Actual); Primary Completion 2016-10-05 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Piccioni, MD, PhD, Principal Investigator — University of California Medical Center
Locations (1):
- The Rebecca and John Moores UCSD Cancer Center, La Jolla, California, United States

REFERENCES:
- [Derived] Piccioni D, Juarez TM, Kesari SL, Rose L, Nomura N, Kesari S. Phase II trial of nilotinib in PDGFR-alpha-enriched recurrent high-grade gliomas. Neurooncol Adv. 2025 Jul 10;7(1):vdaf150. doi: 10.1093/noajnl/vdaf150. eCollection 2025 Jan-Dec. PMID 40709015

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 38 people were enrolled in the study and 34 were treated with study drug. When patients came off treatment they moved into survival follow up.
Period: Overall Study
Arm/Group | Nilotinib
Started (Patients who signed study consent) | 38
Screen Fail | 4
Treated With Study Drug | 34
Completed (Patients who were still on study at the time of closure) | 2
Not Completed | 36
Not completed — disease progression | 31
Not completed — Withdrawal by Subject | 1
Not completed — Screen Fail | 4

BASELINE CHARACTERISTICS:
Arm/Group | Nilotinib
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Had 6-month Progression-free Survival.
Description: Progression was defined by McDonald Criteria: A 25% increase in the sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease) using the same techniques as baseline, OR clear worsening of any evaluable disease, OR appearance of any new lesion/site, OR clear clinical worsening OR failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: 6 months
Population: 38 patients were enrolled, but only 34 were treated
Measure: Count of Participants; unit: Participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 34
Participants | 3

2. Secondary Outcome: Overall Response Rate
Description: How many patients who had decrease in tumor size or complete disappearance of tumor.
Time Frame: 5 years
Population: 38 patients enrolled, but only 34 received study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 34
Participants | 1

ADVERSE EVENTS:
Time Frame: 8 years
Description: used clinicaltrials.gov definitions
Arm/Group | Nilotinib
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 3/34
Other Adverse Events (participants affected / at risk) | 24/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=34)
Musculoskeletal tissue disorder-other: Muscle Spasm (Musculoskeletal and connective tissue disorders) | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=34)
Alkaline Phosphatase Increased (Investigations) | 2
ALT Increase (Investigations) | 2
Anemia (Blood and lymphatic system disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
AST Increased (Investigations) | 2
Confusion (Psychiatric disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 2
Headache (Nervous system disorders) | 3
Fatigue (Investigations) | 5
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Insomnia (Psychiatric disorders) | 2
Localized Edema (General disorders) | 3
Rash Acneiform (Skin and subcutaneous tissue disorders) | 2
Seizure (Nervous system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Pain (General disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes